CLINICAL TRIAL: NCT07002138
Title: The Acceptability of Digital Impression Compared to Conventional Technique in Children - A Randomized Controlled Clinical Trial
Brief Title: The Acceptability of Digital Impression Compared to Conventional Technique in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beirut Arab University (Other)
Responsible Party: Principal Investigator, Hind Tabbal, Clinical Professor, Beirut Arab University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2023-H-0139-D-M-0578
Record Dates: First submitted 2025-05-17; First posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Dental Anxiety; Gagging; Dental Impression Techniques; Pediatric Dentistry
Keywords: intraoral scanners; pediatric dentistry; gag reflex; alginate impressions; children preference; parents preference
MeSH Terms: conditions — Gagging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence A: Conventional First, then Digital (Experimental): Participants in this group receive a conventional alginate impression first (Hydrogum 5, Zhermack), followed by a digital intraoral scan (medit i700) (after a 14-21 day washout period).
  Interventions: Device: Digital Dental Impression; Procedure: Conventional Dental Impression
- Sequence B: Digital First, then Conventional (Experimental): Participants in this group receive a digital intraoral scan first (medit i700), followed by a conventional alginate impression (Hydrogum 5, Zhermack) after a 14-21 day washout period.
  Interventions: Device: Digital Dental Impression; Procedure: Conventional Dental Impression

INTERVENTIONS:
Device: Digital Dental Impression — Digital dental impressions were performed using the Medit i700 intraoral scanner (Medit, Seoul, South Korea). The scanner utilizes 3D-in-motion video technology with UV-C and LED light sources and adaptive anti-fogging. Scans were taken of both upper and lower arches following manufacturer-recommended protocols. Two tip sizes were used (normal and small), and scanning included occlusal, lingual, and buccal surfaces. Moisture control was maintained with cheek retractors and saliva ejectors. Impression time was recorded using a chronometer. This procedure was used to evaluate patient comfort, anxiety, and preference.
  Other Names: Intraoral scan
Procedure: Conventional Dental Impression — Conventional impressions were taken using extra-fast setting flavored alginate (Hydrogum 5, Zhermack SpA, Italy) for both upper and lower arches. The impression material was manually mixed according to the manufacturer's instructions and applied using standard perforated plastic trays suitable for pediatric arches. Children were seated upright, and the impression sequence followed lower arch first, then upper arch. Comfort was evaluated using VAS scores and anxiety using the Venham Clinical Anxiety Scale (VCAS). The procedure was timed with a chronometer.
  Other Names: Alginate impression

SUMMARY:
This randomized crossover clinical trial aims to evaluate the acceptability of digital intraoral impressions compared to conventional alginate impressions in children aged 6 to 11 years. The study will assess patient comfort, anxiety, time efficiency, and preference using validated tools. A total of 40 children who require dental impressions for orthodontic or prosthetic treatment will be enrolled and randomly assigned to receive both impression techniques in alternating order, with a washout period of 14-21 days between sessions. Data collection includes Visual Analog Scale (VAS) scores for comfort and gag reflex, Venham's Clinical Anxiety Scale for anxiety assessment, and comparative questionnaires for both patients and parents. The study aims to determine whether digital impressions offer a more acceptable and less distressing alternative for pediatric patients in clinical dental settings.

DETAILED DESCRIPTION:
This randomized crossover clinical trial aims to evaluate and compare the acceptability, comfort, time efficiency, and anxiety levels associated with digital intraoral impressions versus conventional alginate impressions in children aged 6 to 11 years. Dental impressions are essential in pediatric treatment planning, yet conventional alginate techniques are often poorly tolerated by children due to discomfort, taste, gagging, and procedural anxiety. Advances in digital dentistry, particularly intraoral scanners (IOS), provide a less invasive alternative with potential to enhance patient cooperation and improve the overall experience. Despite their growing use in adult patients, evidence regarding children's acceptance of intraoral scanning remains limited, particularly in the Middle East.

This study will be conducted at the Pediatric Dentistry Department of Beirut Arab University over a four-month period and will involve 40 pediatric patients who require dental impressions for fixed or removable appliances. A 1:1 randomization process will assign participants to one of two sequences: Group 1 will receive a digital impression first, followed by a conventional impression after a 14-21 day washout period; Group 2 will receive the procedures in reverse order. All procedures will be performed by a single calibrated operator.

Digital impressions will be made using the Medit i700 intraoral scanner, which allows 3D image acquisition without physical materials or trays. The scanning process includes drying the teeth and capturing occlusal, lingual, and buccal surfaces. Conventional impressions will be obtained using Hydrogum 5 alginate, involving tray selection, alginate mixing, and taking maxillary and mandibular impressions, followed by disinfection.

To assess acceptability and experience, several outcome measures will be recorded. Patient comfort and specific sensory responses will be measured using a Visual Analog Scale (VAS), where children will rate domains such as general feeling, breathing difficulty, taste or smell discomfort, thermal discomfort (heat/cold), gag reflex, and pain. Operator-assessed anxiety levels will be scored using the Venham's Clinical Anxiety Scale (VCAS), ranging from 0 (no anxiety) to 5 (severe anxiety). Total procedure time will be recorded using a digital stopwatch, beginning at tray or scanner insertion and ending at procedure completion. After both procedures, a structured comparative questionnaire will be administered to children, their parents, and the operator to assess perceived comfort, ease, duration, and preference.

Additionally, the operator's subjective perception of difficulty, applicability, and preference for each method will be documented. Intra-examiner reliability for digital scanning will be evaluated using repeated scans of 10 cases at a 48-hour interval, with agreement assessed via Cohen's Kappa statistic.

Statistical analysis will be conducted using SPSS version 26. Normality testing will guide the use of parametric or non-parametric tests (e.g., paired t-test or Wilcoxon signed-rank test), with a significance level set at α = 0.05. Descriptive statistics will be presented for baseline demographic data.

The study has been approved by the Ethics Committee of Beirut Arab University (Protocol ID: 2023-H-0139-D-M-0578). Informed consent will be obtained from parents or legal guardians before participation, and confidentiality will be strictly maintained. Participants will not incur costs or receive compensation.

By comparing these two impression methods in terms of comfort, anxiety, and feasibility, this study aims to generate original data relevant to pediatric dentistry and digital workflows. The findings may inform best practices and encourage the adoption of child-friendly technologies in clinical dental care.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6-11 years
* In need for the fabrication of fixed or removable appliance
* Having gagging problem based on the Classification of Gagging Problem scale starting from G1 to G5. (Saita et al., 2013) Where G1 is Normal Gagging: Normal gagging but not desensitized (controlled by the patient). The patient can withstand a full mouth examination with a dental mirror and a basic periodontal examination G2 is Mild gagging : Gagging when probe was used in a basic periodontal examination G3 is Moderate gagging: Gagging when examining molar teeth with a mirror G4 is Severe gagging: Gagging when examination of anterior teeth with a mirror G5 is Very severe gagging: Gagging at the moment when the dental mirror is inserted

Exclusion Criteria:

* Having a previous experience with any type of dental impressions.
* Having any systemic diseases or mental disorders.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-05-17 (Actual); Study Completion 2024-05-17 (Actual)

PRIMARY OUTCOMES:
Comparison of patient comfort during digital and conventional methods | Assessed immediately following each impression procedure during the same clinical visit
  Child comfort level during each impression was recorded using the Visual Analogue Scale (VAS), a 6-point questionnaire 10 cm VAS where "10" represented maximum complaint whereas the value "0" meant no discomfort and better outcome. Scores were documented by the operator and analyzed across impression type, cooperation level, and gag reflex severity.
Duration of digital versus conventional dental impressions | Assessed immediately following each impression procedure during the same clinical visit
  Time (in seconds) required to complete each impression was measured using a chronometer. Timing included preparation and execution phases. Durations for digital (Medit i700) and conventional (Hydrogum 5) impressions were compared across age groups, gag reflex severity, scanner tip size, and cooperation levels

SECONDARY OUTCOMES:
Comparison of child anxiety levels during digital and conventional impressions | Assessed immediately following each impression procedure during the same clinical visit.
  Child anxiety during each impression was recorded using the Venham Clinical Anxiety Scale (VCAS), a 6-point behavioral assessment, where 0 represent no anxiety and 5 presents the maximum anxiety and worst outcome. Scores were documented by the operator and analyzed across impression type, cooperation level, and gag reflex severity.
Comparison of patient and caregiver preferences for digital versus conventional impressions | Assessed immediately after digital procedure during the same clinical visit.
  Children and their caregivers completed structured questionnaires after both impression procedures. Preferences were recorded for future use, perceived comfort, and overall experience with digital (Medit i700) versus conventional alginate (Hydrogum 5) impressions. Preferences were analyzed separately for impressions of the upper and lower arches.
Comparison of operator perception of difficulty and applicability of digital versus conventional impressions | Assessed immediately after both impressions were completed for each participant during the same clinical session.
  The operator completed a structured questionnaire after both impression procedures for each participant. The questionnaire assessed perceived level of difficulty, ease of application, and overall preference between the digital (Medit i700) and conventional (Hydrogum 5) methods. Results were analyzed to evaluate workflow challenges and usability from the clinician's perspective.

CONTACTS AND LOCATIONS:
Overall Officials: Associate Professor Ahmad Tarabaih, Associate Professor Ahmad, Study Director — Beirut Arab University
Locations (1):
- The Pediatric Dental clinics of the Faculty of Dentistry at Beirut Arab University, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No